CLINICAL TRIAL: NCT03236155
Title: Comparing Opioid Prescription Patterns in Total Joint Arthroplasty Patients: A Randomized Controlled Trial
Brief Title: Comparing Opioid Prescription Patterns in Total Joint Arthroplasty Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Attending Physician, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17030306
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Pain
Keywords: Opioids
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 prescription (Active Comparator): Receives 90 pills in single prescription at discharge from hospital
  Interventions: Drug: opioid pain pills
- 3 prescriptions (Active Comparator): Receives 30 pill prescription at discharge from hospital. Two refills available if requested.
  Interventions: Drug: opioid pain pills

INTERVENTIONS:
Drug: opioid pain pills — patient will receive their pain pill prescription

SUMMARY:
The United States constitutes <5% of the world's population but over 80% of the opioid supply and 99% of the hydrocodone supply. In 2014, there were 18,893 deaths from prescription drug overdose, and orthopaedic surgeons are the third highest prescribing physicians for opioids. Surgeons often prescribe opioids to minimize postoperative pain and to reduce the likelihood of readmission for pain. Available data suggests that orthopaedic surgeons are the most likely physicians to prescribe opioids to Medicare patients, whose opioid prescriptions are over 7 times more likely to come from an orthopaedic surgeon than another type of physician, but orthopaedic surgeons also had the highest readmission rate for post-operative pain. Many studies have investigated the utilization of opioids after surgery to assess surgeon's tendencies to overprescribe, demographics of those likely to overuse, and adverse events of opioid abusers.

The primary purpose of this randomized controlled trial is to determine whether prescribing fewer opioid pills per prescription reduces the total amount of opioids taken, even while allowing equal total opioid availability via increased frequency of prescription availability.

DETAILED DESCRIPTION:
A recent paper by Kim et al prospectively investigated opioid utilization after upper extremity surgery. This study (n=1,416) showed an opioid utilization rate of just 34%, taking an average 8.1 pills out of 24 prescribed. Patients age 30-39, those having joint procedures, upper extremity/shoulder surgery, or self-pay/Medicaid insurance were all far more likely to overuse opioids. The study concluded that their surgeons prescribed 3 times the required opioid following surgery and gave recommendations for opioid distribution based on location, procedure type, and patient risk factors. This study's identification of over prescription is congruent with a study completed by Bates et al that showed 67% of patients had a surplus of medications, with 92% not receiving proper medication disposal instructions.

Other recent literature has attempted to risk stratify patients who are more likely to abuse prescription opioids. Morris et al identified various risk factors including: family history of substance abuse, nicotine dependency, age <45, psychiatric disorders, and lower level of education. These risk factors are associated with aberrant behaviors (non-compliance, early refill request, "lost or stolen" medication), which should raise concerns for any provider prescribing opioids.

Studies have shown that patients who are on chronic opioid therapy before surgery have worse outcomes. Nicholas Bedard et al compared chronic opioids users (n= 35,068) versus those who were opioid-naïve at the time of total knee arthroplasty (TKA) and found the opioid group had more opioid scripts filled per patient at discharge as well as at 3, 6, and 9 months (0.63 scripts/patient vs. 1.2 scripts/patient, p<0.05). These patients also had a higher Charlson Comorbidity Index (p<0.05) and higher rates of respiratory failure, acute kidney failure, pneumonia, all post-operative infections, and infections requiring return to the OR. The study concluded patients should have their opioid consumption controlled during the pre-operative and peri-operative period.

In addition to the complications of opioid medications experienced by orthopaedic patients, a recent nationwide retrospective analysis presents an unintended yet severe problem associated with opioid prescriptions. The incidence of pediatric hospitalizations for opioid toxicity nearly tripled from 1997 to 2012. The over-prescription of opioids creates a readily available source for accidental ingestion by younger children and for intentional opioid overdose by older pediatric/adolescent patients. In fact, a family member's leftover pills have been described as the number one source for pediatric opioid overdose. Moreover, the Center for Disease Control reported that in 2015 the U.S. saw its highest incidence of opioid-related death.9 Given the frequency and severity of opioid diversion and misuse, orthopaedic surgeons should consider the best methods for controlling patients postoperative pain and also avoid facilitating opiate misuse, whether by orthopaedic patients or other community members. With this goal in mind, our study will investigate regimens for effective postoperative pain control that also minimize the total amount of opioids prescribed.

ELIGIBILITY:
Inclusion Criteria:

* any patient > 18 years of age scheduled for primary total hip or knee arthroplasty who is not consuming opioids during the 4 weeks prior to surgery

Exclusion Criteria:

* patients consuming opioids during the 4 weeks prior to surgery
* patients who are allergic to oxycodone or refuse to take oxycodone
* patients with a history of opioid dependence or illegal or "off-label" opioid use
* patients undergoing a revision total knee or total hip arthroplasty
* any patient less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim N, Matzon JL, Abboudi J, Jones C, Kirkpatrick W, Leinberry CF, Liss FE, Lutsky KF, Wang ML, Maltenfort M, Ilyas AM. A Prospective Evaluation of Opioid Utilization After Upper-Extremity Surgical Procedures: Identifying Consumption Patterns and Determining Prescribing Guidelines. J Bone Joint Surg Am. 2016 Oct 19;98(20):e89. doi: 10.2106/JBJS.15.00614. PMID 27869630
- [Background] Opioid Addiction 2016 Facts & Figures. American Society of Addiction Medicine. Retrieved from: http://www.asam.org/docs/default-source/advocacy/opioidaddiction-disease-facts-figures.pdf
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Bedard Nicholas, Callaghan John, Pugely Andrew, Martin Christopher, Duchman Kyle, Westermann Robert, Gao Yubo. Pre-Opioid Use: Is There an Association with Outcomes Following Total Knee Arthroplasty? In: American Academy of Orthopaedic Surgeons 2016 Annual Meeting; 2016 Mar 1-5; Orlando, FL. Presentation nr P161
- [Background] Bates C, Laciak R, Southwick A, Bishoff J. Overprescription of postoperative narcotics: a look at postoperative pain medication delivery, consumption and disposal in urological practice. J Urol. 2011 Feb;185(2):551-5. doi: 10.1016/j.juro.2010.09.088. Epub 2010 Dec 18. PMID 21168869
- [Background] Opioid Use, Misuse, and Abuse in Orthopaedic Practice. American Academy of Orthopaedic Surgeons. October 2015. Retrieved from: http://www.aaos.org/uploadedFiles/PreProduction/About/Opinion_Statements/adv istmt/1045%20Opioid%20Use,%20Misuse,%20and%20Abuse%20in%20Practice .pdf
- [Background] Gaither JR, Leventhal JM, Ryan SA, Camenga DR. National Trends in Hospitalizations for Opioid Poisonings Among Children and Adolescents, 1997 to 2012. JAMA Pediatr. 2016 Dec 1;170(12):1195-1201. doi: 10.1001/jamapediatrics.2016.2154. PMID 27802492
- [Background] Moreno MA. Page for patients. The misuse of prescription pain medicine among children and teens. JAMA Pediatr. 2015 May;169(5):512. doi: 10.1001/jamapediatrics.2014.2128. No abstract available. PMID 25938654
- [Background] Retrieved on 12/9/16 from: https://www.whitehouse.gov/the-pressoffice/2016/12/08/continued-rise-opioid-overdose-deaths-2015-shows-urgentneed-treatment
- [Background] Della Valle CJ, Dittle E, Moric M, Sporer SM, Buvanendran A. A prospective randomized trial of mini-incision posterior and two-incision total hip arthroplasty. Clin Orthop Relat Res. 2010 Dec;468(12):3348-54. doi: 10.1007/s11999-010-1491-5. Epub 2010 Jul 29. PMID 20668969

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Prescription | 3 Prescriptions
Started | 143 | 161
Completed | 143 | 161
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Minimum Age: 18 Years Maximum Age: none Sex: All Gender Based: No Ethnicity Based: no
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Prescription | 3 Prescriptions | Total
Number analyzed (Participants) | 143 | 161 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 83 | 153
  >=65 years | 73 | 78 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 89 | 164
  Male | 68 | 72 | 140
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 143 | 161 | 304

OUTCOME MEASURES:

1. Primary Outcome: Morphine Milligram Equivalents (MME) of Oxycodone Tablets Taken by Patient
Description: Self-reported by patient, we are asking for the number of Oxycodone taken by patients (5mg doses). This will be verified with patient bringing their pill bottle in and counted by a study investigator.
Time Frame: 30 days
Population: Opioid naive patients undergoing THA or TKA between August 2017 and April 2018 and Morphine Milligram Equivalents (MME) of Oxycodone Tablets Taken by Patient
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Groups:
- 90 (5mg OxyIR) Pills Prescribed: Receives 90 pills in single prescription at discharge from hospital
  opioid pain pills: patient will receive their pain pill prescription
- 30 (5mg OxyIR) Pills Prescribed: Receives 30 pill prescription at discharge from hospital. Two refills available
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Pills Prescribed
Number analyzed (Participants) | 143 | 161
Morphine Milligram Equivalents (MME) | 1089.7 (536.4) | 777.1 (414.2)

2. Secondary Outcome: Postoperative Patient Reported Outcomes of Opioid naïve Patients Undergoing THA or TKA Between August 2017 and April 2018
Description: Postoperative total hip and total knee arthroplasty patient reported outcomes at 90 days (All reported as scores on a scale, ranges below.). For hips: Hip Disability and Osteoarthritis Outcome Score Joint Replacement (Hoos Jr), for knees: Knee Injury and Osteoarthritis Outcome Score, Joint Replacement, (Koos Jr), additionally, all will complete the Veterans Rand-12 outcome (VR-12). All outcomes, closer to 100 are better outcomes.
  HOOS, JR: Questions coded 0 - 4 points, none - extreme pain, scored by summing responses (range 0-24), convert to t-score. Answer ranges 0 - 100 (0 - total hip disability, 100 -perfect hip health).
  KOOS, Jr: Same but for Knees VR-12: Assesses physical functioning, physical/ mental limitations. Scored as summary of mental/physical, measure in standard deviations out of 100 points, where a score of 100 shows a patient's health functioning physically and mentally at their their best, zero represents a worse outcome.
Time Frame: 90 days post operative (higher values represent better functioning total hip or total knee replacements).
Population: Scores closer to 100 are considered better outcomes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 30 (5mg OxyIR) Pills Prescribed: Receives 30 pill prescription at discharge from hospital. Two refills available if requested.
  opioid pain pills: patient will receive their pain pill prescription
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Pills Prescribed
Number analyzed (Participants) | 143 | 161
score on a scale
  Postop Koos Jr | 65.9 (9.9) | 65.0 (11.7)
  Postop Hoos Jr | 73.5 (13.8) | 73.7 (12.3)
  Postop VR-12 | 93.2 (14.7) | 92.1 (14.3)

3. Secondary Outcome: Complications
Description: Complications will be recorded as follows post-operatively for 90 days following surgery; any patient that has a DVT/Pulmonary embolism, any return to the operating room within 90-days, any re-admission to the hospital within 90-days, Any report of superficial infection, any report of deep infection, a periprosthetic fracture of the joint replaced, cerebrovascular accident or transient ischemic attack, report of dislocation, or patients who report opioid withdrawal.
Time Frame: 90 days from time of surgery
Population: 304 opioid naive patients undergoing total hip or total knee arthroplasties
Measure: Count of Participants; unit: Participants
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Pills Prescribed
Number analyzed (Participants) | 143 | 161
Participants | 0 | 0

4. Secondary Outcome: Compliance
Description: This will be done as monitored through the Illinois prescription monitoring program, collecting data on each patient enrolled to be sure that patients do not receive additional narcotic prescriptions beyond what is provided to them as part of the study.
Time Frame: 90 days
Measure: Number; unit: Number of Compliant Participants
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Pills Prescribed
Number analyzed (Participants) | 143 | 161
Number of Compliant Participants | 143 | 161

5. Secondary Outcome: Preoperative Patient Reported Outcomes
Description: Utilizing Preop Koos Jr, Preop Hoos Jr, and Pre operative VR-12, all subjects will be asked to provide a pre-operative patient reported outcome to compare to post-operative patient reported outcomes. All reported as scores on a scale, ranges below.
  HOOS, JR: Questions coded 0 to 4 points, none to extreme pain, scored by summing responses (range of 0-24), convert to interval score ranges 0 to 100 (0 - total hip disability, 100 -perfect hip health).
  KOOS, Jr: Same but for Knees VR-12: Assesses physical functioning, physical/ mental limitations. Scored as summary of mental and physical, measure in standard deviations. The scale range is 0 to 100, where a score of 100 represents the best physical and mental health and zero is the worst outcome.
Time Frame: 10 days prior to surgery (higher values represent better functioning total hip or total knee replacements).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Pills Prescribed
Number analyzed (Participants) | 143 | 161
score on a scale
  Preop Koos Jr | 49.3 (12.5) | 51.5 (13.6)
  Preop Hoos Jr | 53.2 (16.3) | 50.7 (15.9)
  Preop VR-12 | 90.8 (14.6) | 89.1 (16.1)

6. Secondary Outcome: Postoperative Outpatient Pain Scores
Description: Utilizing the defense & veterans pain rating scale, patients enrolled will be asked at multiple time points after surgery regarding their pain. This is a pain assessment tool, using numerical rating scale, 0 (no pain), 1, 2, and 3 (mild), 4, 5, and 6 (moderate), 7, 8, and 9 (severe) to 10 (worst pain possible). The higher the score, the more pain.
Time Frame: Days 1-3, 1 week, 2 weeks, and 3-4 weeks post discharge from surgery
Population: 304 opioid naïve patients undergoing THA or TKA, assessed daily from time of surgery to discharge from hospital (1 days - 4 weeks), Reported at 1-3 days, 1 week after surgery, 2 weeks after surgery, and 3-4 weeks after surgery (dependent on follow up appointment).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Pills Prescribed
Number analyzed (Participants) | 143 | 161
score on a scale
  Days 1-3 after discharge | 4.0 [0 to 10] | 4.3 [0 to 8.3]
  Week 1 after discharge | 3.9 [0.4 to 10] | 4.1 [0.3 to 7.7]
  Week 2 after discharge | 3.3 [0 to 9.6] | 3.1 [0 to 7.6]
  Weeks 3-4 after discharge | 2.2 [0 to 8.4] | 2.2 [0 to 6.3]

7. Secondary Outcome: Postoperative Inpatient Opioid Utilization
Description: Using the primary outcome of number of opioids taken by the patients while inpatient, those will be converted into morphine equivalents. This was obtained from the hospital chart during the patient's inpatient stay.
Time Frame: from time of surgery to discharge from hospital (1 day - 2 weeks)
Population: 304 opioid naïve patients undergoing THA or TKA between August 2017 and April 2018
Measure: Mean (Standard Deviation); unit: Morphine Equivalent while inpatient
Groups:
- 30 (5 mg OxyIR) Pills Prescribed: Receives 30 pill prescription at discharge from hospital. Two refills available if requested.
  opioid pain pills: patient will receive their pain pill prescription
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5 mg OxyIR) Pills Prescribed
Number analyzed (Participants) | 143 | 161
Morphine Equivalent while inpatient | 64.6 (38.9) | 72.2 (55.9)

8. Secondary Outcome: Postoperative Inpatient Pain Scores
Description: Using a Defense and Veterans Pain Rating scale, patients were asked from date of surgery to the date of discharge for daily inpatient pain scores. This is a pain assessment tool, using numerical rating scale, 0 (no pain), 1, 2, and 3 (mild), 4, 5, and 6 (moderate), 7, 8, and 9 (severe) to 10 (worst pain possible). The higher the score, the more pain.
Time Frame: assessed daily from time of surgery to discharge from hospital (1 days - 2 weeks), Day 14 scores reported
Population: 304 opioid naïve patients undergoing THA or TKA between August 2017 and April 2018
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- 90 (5mg OxyIR) Prescribed: Receives 90 pills in single prescription at discharge from hospital
  opioid pain pills: patient will receive their pain pill prescription
- 30 (5mg OxyIR) Prescribed: Receives 30 pill prescription at discharge from hospital
  opioid pain pills: patient will receive their pain pill prescription
Arm/Group | 90 (5mg OxyIR) Prescribed | 30 (5mg OxyIR) Prescribed
Number analyzed (Participants) | 143 | 161
score on a scale | 4 [0 to 8.7] | 4.5 [0 to 10]

9. Secondary Outcome: Number of Tablets Received From Pharmacy That Went Unused
Description: 304 opioid naïve patients undergoing THA or TKA between August 2017 and April 2018, reporting number of pills not used
  Illinois prescription monitoring program- utilized to confirm no other physician prescribed opiates to the participating patients. They were asked at each visit regarding unused medications and brought to the office to properly dispose.
Time Frame: 90 days
Measure: Median (Full Range); unit: Unused pills
Groups:
- 30 (5mg OxyIR) Prescribed: Receives 30 pill prescription at discharge from hospital. Two refills available if requested.
  opioid pain pills: patient will receive their pain pill prescription
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Prescribed
Number analyzed (Participants) | 143 | 161
Unused pills | 73 [0 to 90] | 15 [0 to 30]

ADVERSE EVENTS:
Time Frame: 304 opioid naïve patients following their THA or TKA for 90 days, for surgeries between August 2017 and April 2018 agreed to participate and were randomized to two groups: 30 or 90 5-mg oxycodone immediate release (OxyIR) pills after discharge.
Description: no difference in definition.
Arm/Group | 90 (5mg OxyIR) Pills Prescribed | 30 (5mg OxyIR) Pills Prescribed
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/161
Other Adverse Events (participants affected / at risk) | 0/143 | 0/161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03236155/Prot_SAP_002.pdf